CLINICAL TRIAL: NCT06906965
Title: Impact of the Imera Carob Cultivar in Postprandial Glycemia
Brief Title: Effect of the Imera Cultivar Carob in Postprandial Glycemia
Acronym: IMERACAROBGLUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C. Kaliora, Professor, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CAROB_GLUCOSE_147; 016713 (Other Grant/Funding Number: Hellenic Foundation for Research and Innovation)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Postprandial Glucose Regulation
Keywords: postprandial glucose; glucose regulation; carob; carob powder; postprandial insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carob beverage (Experimental): The participants consumed a carob beverage prepared with 30 g of Imera cultivar carob powder dissolved in water
  Interventions: Other: Carob beverage
- Sucrose beverage (Active Comparator): The participants consumed a sucrose beverage made containing 14 g of sugar, matched to the sugar concentration of the experimental beverage
  Interventions: Other: Sucrose beverage

INTERVENTIONS:
Other: Carob beverage — The participants consumed a carob beverage made with 30gr of Imera carob cultivar powder in water
  Arms: Carob beverage
Other: Sucrose beverage — The participants consumed a sucrose beverage made with 14gr of sugar in alike concentration with sugars in the experimental beverage
  Arms: Sucrose beverage

SUMMARY:
An acute randomized crossover study on the effect of a carob beverage on postprandial glycemic response

DETAILED DESCRIPTION:
This is an acute randomized crossover study on the effect of an Imera cultivar carob beverage on postprandial glycemic response in healthy individuals as opposed to sucrose-based beverage containing sugar in alike concentration

ELIGIBILITY:
Inclusion Criteria:

* healthy male adults of normal body fat mass

Exclusion Criteria:

* obesity (according to body fat mass), type 1 Diabetes, hypertension and other cardiovascular diseases, thyroid disorder, liver, kidney, gastrointestinal disease, mental illness, use of nutraceutical supplements or natural products for weight loss and the background of dietitian/nutritionist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | 3 hours
  Changes in glucose levels after the consumption of the beverage

SECONDARY OUTCOMES:
Postprandial insulin | 3 hours
  Changes in insulin levels after consuming the beverage

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition and Dietetics, HarokopioUniversity of Athens, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: No